CLINICAL TRIAL: NCT01703455
Title: Sorafenib in Recurrent and/or Metastatic Salivary Gland Carcinomas: Phase II Study
Brief Title: Activity of Sorafenib in Salivary Gland Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Lisa Licitra, Prof. MD, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INT29/10
Record Dates: First submitted 2012-04-06; First posted 2012-10-10 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Salivary Gland Cancer
Keywords: Salivary gland metastatic recurrent disease clinical trial
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib 400 mg twice daily (Experimental): Sorafenib 400 mg twice daily, on a continuous basis (each morning and evening), in 4 week cycles
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — 400 mg twice daily, on a continuous basis (each morning and evening), in 4 week cycles
  Other Names: Nexavar

SUMMARY:
This is a single agent, prospective, open-label, monocenter, phase II trial of sorafenib in patients with recurrent and/or metastatic salivary gland carcinoma. This trial will be conducted with the primary aim to determine the response rate (CR+PR) according to the RECIST criteria. Response rate according to CHOI criteria, correlation between CHOI criteria and outcome, disease Control Rate (DCR) and acute toxicity will be evaluated as secondary objectives.

DETAILED DESCRIPTION:
This phase II trial was conducted on adult patients with RMSGC. Inclusion criteria were as follows: histologically proven diagnosis of RMSGC; availability of primary tissue (block or formalin fixed paraffin embedded [FFPE] tissue slides); age _18 years; Eastern Cooperative Oncology Group Performance Status (ECOG-PS) 0e1; adequate bone marrow, liver and renal function (haemoglobin >9.0 g/dl; neutrophil count >1500/mm3; platelet count _100,000/ml; total bilirubin <1.5 _ upper limit of normal [ULN]; ALT and AST <2.5 _ ULN and <5 _ ULN for patients with liver metastases; serum creatinine <1.5 _ ULN; alkaline phosphatase <4 _ ULN; PT-INR/PTT <1.5 _ ULN); _1 measurable unidimensional lesion by magnetic resonance imaging (MRI) or computed tomography (CT) scan according to the RECIST 1.1 criteria. Patients with cardiac disease (i.e. congestive heart failure New York Heart Association (NYHA) > 2, cardiac arrhythmia; uncontrolled hypertension) in the six months before study entry were excluded. Previous chemotherapy for metastatic disease was allowed and progression of disease was not required for the enrolment. All patients provided written informed consent. The study was conducted in accordance with Good Clinical Practice guidelines and the Declaration of Helsinki and was approved by the local Ethical Committee (Registry number, NCT01703455). 2.2. Treatment and assessments: Patients received 400 mg of sorafenib orally every 12 h on a continuous basis in 4-week cycles until disease progression and/or unacceptable toxicity. Biochemical and clinical evaluation, and drug safety monitoring according to the Common Terminology Criteria for Adverse Events (CTCAE) v3.0 were performed every 4 weeks. The attribution of adverse events (AEs) to the study drug was judged by the investigators. CT scans were performed every 8 weeks until disease progression. An independent evaluation of radiological response (RECIST and Choi criteria) was performed by two radiologists on anonymised CT scans. Stomatology evaluation was performed at baseline to exclude any sign of osteoradionecrosis. Dose reduction was adopted in cases of clinically significant haematologic or other AEs that were considered related to sorafenib. In such cases, doses were reduced to 400 mg once daily and then to 400 mg every other day. If further reductions were required, patients were withdrawn from the trial. Dose reescalation was not allowed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven relapsed and/or metastatic salivary gland cancer for which potentially curative options such as surgery or radiotherapy are not indicated
* One target lesion measurable by CT-scan or MRI according to RECIST criteria
* Age + 18 years
* ECOG 0 or 1
* Adequate bone marrow, liver and renal function
* Signed written informed consent

Exclusion Criteria:

* Symptomatic metastatic brain or meningeal tumors
* History of cardiac disease such as congestive heart failure>NYHA class 2
* Active CAD
* Cardiac arrhythmias requiring anti-arrhythmic therapy or uncontrolled hypertension
* Pregnant or breast-feeding patient
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Patients unable to swallow oral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Objective response | 8 weeks
  Response Rate according to RECIST criteria. Response will be evaluated every 2 months.

SECONDARY OUTCOMES:
response rate according to CHOI criteria | 8 weeks
  assessment of tumor response according to CHOI criteria
correlation between CHOI criteria and outcome | one year
  correlation between CHOI criteria and survival (OS and PFS)

OTHER OUTCOMES:
adverse events | 4 weeks
  number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, MD, Prof, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- IRCCS Istituto Nazionale Tumori, Milan, Italy